CLINICAL TRIAL: NCT05597800
Title: A Phase 2, Multicenter, Open Label, Clinical Trial Evaluating Safety and Activity of Nivolumab/Ipilimumab and Chemotherapy Combination in Advanced NSCLC Patients With HIV, HBV, HCV and Post-acute Sequelae of SARS-CoV2 Infection (PASC).
Brief Title: Nivolumab/Ipilimumab and Chemotherapy Combination in Advanced NSCLC Patients With HIV, HBV, HCV and Long Covid Syndrome
Acronym: LUNGVIR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Lorenzo Belluomini, Principal Investigator, Medical Oncologist, Universita di Verona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-002313-41; 2022-002313-41 (EudraCT Number)
Record Dates: First submitted 2022-10-21; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: NSCLC Stage IV; HIV; HBV; HCV; Long COVID
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Post-Acute COVID-19 Syndrome | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Study type: Phase 2 - Interventional Trial Study drugs: nivolumab and ipilimumab Cohort A: HBV and HCV patients Cohort B: HIV patients Cohort C: Long COVID syndrome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A: HBV and HCV patients (Experimental): Participants (≥ 18 years) must have histologically confirmed metastatic or unresectable non-small cell lung cancer (both non-squamous and squamous), without sensitizing EGFR, ALK, ROS1, BRAF and NTRK alterations, with chronic viral infections, such as HBV and HCV in cohort A.
  Squamous histology: carboplatin AUC 6 + paclitaxel 200 mg/m2 Non-squamous histology: carboplatin AUC 5 or 6 + pemetrexed 500 mg/m2 or cisplatin 75 mg/m2 + pemetrexed 500 mg/m2.
  Interventions: Drug: Nivolumab and Ipilimumab
- Cohort B: HIV patients (Experimental): Participants (≥ 18 years) must have histologically confirmed metastatic or unresectable non-small cell lung cancer (both non-squamous and squamous), without sensitizing EGFR, ALK, ROS1, BRAF and NTRK alterations, with chronic viral infections such as HIV in cohort B.
  Squamous histology: carboplatin AUC 6 + paclitaxel 200 mg/m2 Non-squamous histology: carboplatin AUC 5 or 6 + pemetrexed 500 mg/m2 or cisplatin 75 mg/m2 + pemetrexed 500 mg/m2.
  Interventions: Drug: Nivolumab and Ipilimumab
- Cohort C: Long COVID syndrome (Experimental): Participants (≥ 18 years) must have histologically confirmed metastatic or unresectable non-small cell lung cancer (both non-squamous and squamous), without sensitizing EGFR, ALK, ROS1, BRAF and NTRK alterations, with chronic viral infections such as Long Covid syndrome in Cohort C.
  Squamous histology: carboplatin AUC 6 + paclitaxel 200 mg/m2 Non-squamous histology: carboplatin AUC 5 or 6 + pemetrexed 500 mg/m2 or cisplatin 75 mg/m2 + pemetrexed 500 mg/m2.
  Interventions: Drug: Nivolumab and Ipilimumab

INTERVENTIONS:
Drug: Nivolumab and Ipilimumab — Nivolumab will be administered with ipilimumab, plus 2 cycles of histology-based platinum doublet chemotherapy:
  * Squamous histology: carboplatin AUC 6 + paclitaxel 200 mg/m2
  * Non-squamous histology: carboplatin AUC 5 or 6 + pemetrexed 500 mg/m2 or cisplatin 75 mg/m2 + pemetrexed 500 mg/m Dosing: nivolumab 360 mg every 3 weeks + ipilimumab 1 mg/kg every 6 weeks (up to maximum 2 years) + histology-based, platinum doublet chemotherapy (every 3 weeks for two cycles).
  Other Names: Opdivo and Yervoy

SUMMARY:
Study type: Phase 2 - Interventional Trial Number of patients to be enrolled: 105 Participating countries: Italy Study drugs: nivolumab and ipilimumab Cohort A: HBV and HCV patients Cohort B: HIV patients Cohort C: Long COVID syndrome The stratification factors are HBV/HCV positive (cohort A), HIV positive (cohort B), patients with Long Covid syndrome (Cohort C), histology (squamous vs non-squamous histology), and gender (male vs female).

DETAILED DESCRIPTION:
Participants (≥ 18 years) must have histologically confirmed metastatic or unresectable non-small cell lung cancer (both non-squamous and squamous), without sensitizing EGFR, ALK, ROS1, BRAF and NTRK alterations, with chronic viral infections, such as HBV and HCV in cohort A and HIV in cohort B and with Long Covid syndrome in Cohort C.

The study is a multicenter, open-label trial designed according to Bryant and Day and including 1) a screening phase to establish study eligibility, 2) an open-label treatment phase, in which patients will receive nivolumab plus ipilimumab in combination with histology-based chemotherapy (2 induction cycles) to ascertain its safety, defined as incidence of grade 3 or 4 (G3/4) treatment-related adverse events (TRAEs) and activity, 3) and a follow-up phase to monitor survival status and subsequent therapies.

In detail, the study includes:

1. A screening phase to establish study eligibility (including, for example, the availability of tumour tissue for molecular analyses) and document baseline assessments.
2. An open-label treatment phase, in which patients will be treated with 2 cycles of chemotherapy and nivolumab plus ipilimumab until disease progression, unacceptable toxicity or for a maximum of 2 years. Upon disease progression or completion of trial treatment, further therapy will be at the discretion of the treating physician.
3. A follow-up phase, to monitor safety, survival status and subsequent therapies.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed diagnosis of metastatic or unresectable NSCLC;
* No sensitizing EGFR, ALK, ROS1, BRAF and NTRK alterations;
* Eastern Cooperative Oncology Group (ECOG) score 0-1 (physically able to carry out light housework or office work through to being fully active as they were before cancer);
* No prior systemic anticancer therapy;
* Tissue or Programmed death-ligand 1 (PD-L1) results available;
* HIV-1 or HIV-2 chronic infection, defined as i) a positive HIV 1-2 western blot or other FDA/CE approved HIV confirmatory test (regardless the results of the HIV 1-2 screening test used [2nd, 3rd, 4th generation tests, rapid tests or laboratory tests (i.e., ELISA, EIA, CLIA, etc.)], ii) the referring physician's written record that HIV infection was documented, with supporting information on the participant's relevant medical history and/or current antiretroviral treatment for HIV infection;
* Only subjects with chronic or resolved HBV infections might be eligible. Chronic HBV infections is defined as: the persistence of HBsAg positivity for more than 6 months (regardless HBeAg result, HBV-DNA level and the presence of liver necroinflammation). Resolved HBV infection is defined by: the absence of liver inflammation (clinically and laboratory), HBsAg negativity and HBsAb (anti-HBs antibodies) and HBcAb (anti-HBc IgG) positive result;
* Only subjects with resolved HCV infections might be eligible. Subjects with a newly diagnosed chronic HCV infection (defined as: positive HCV antibodies + detectable HCV-RNA) should be treated for HCV infection before enrollment. Acute HCV infection [defined as a positive HCV-RNA and i) a negative serological HCV assay (HCV-Ab) or ii) a positive serological HCV assay (HCV-Ab) with a negative test 6 months earlier] cannot be enrolled in the study.
* Patients with past HCV infection, with no evidence of chronic infection (i.e., anti-HCV antibody positivity, HCV-RNA negativity) should be excluded;
* Patients with confirmed Long Covid syndrome or PASC defined, as suggest by World Health Organization (WHO), as "condition occurs in individuals with a history of probable or confirmed SARS CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms and that last for at least 2 months and cannot be explained by an alternative diagnosis". This condition must be present at enrollment;
* Participants must have a nasopharyngeal swab positive for Sars-Cov2 within 12 months before enrolment;
* Participants must be either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to first treatment;
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam; scans must have been performed within 4 weeks prior to registration.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug;
* Ability to understand and to sign a written informed consent document.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) score ≥2;
* Untreated symptomatic brain metastases or leptomeningeal metastases;
* Another active concomitant malignancy;
* Active, known or suspected, autoimmune disease;
* Active HBV or HCV infection, presence of any infectious disease requiring specific treatment.
* Active Sars-Cov2 infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Safety, defined as onset of grade 3 or 4 (G3/4) treatment-related adverse events (TRAEs), assessed by the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 5. | 3 years
  The primary objectives of the study are safety, defined as onset of grade 3 or 4 (G3/4) treatment-related adverse events (TRAEs), assessed by the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 5.
Objective Response Rate (ORR) measured as for RECIST 1.1 criteria | 3 years
  Activity in terms of objective response rate (ORR) of nivolumab plus ipilimumab in combination with platinum-based chemotherapy (2 cycles) in first-line advanced NSCLC patients with chronic viral infections.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  Overall survival (OS) is defined as the time between the date of the randomization date and the date of death due to any cause. OS will be censored on the last date a participant was known to be alive.
Progression-free survival (PFS) | 3 years
  Progression free survival (PFS), according to response evaluation criteria in solid tumors (RECIST) 1.1 as assessed by local investigators, is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD is defined as a ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum in study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Duration of response (DOR) | 3 years
  Duration of response (DOR) is defined as the time from date of first documentation of confirmed response (CR or PR) to date of first documentation of progression or symptomatic deterioration, or death due to any cause among patients who achieve, assessed at 6 and 12 months.

OTHER OUTCOMES:
Exploratory objectives | 4 years
  The exploratory analyses include the evaluation of absolute CD4+, CD4/CD8, HIV viral load changes only in cohort B. In cohort A, HBV variables: HBsAg, HBeAg, HBsAb, HBcAb tot e IgM, HBeAb, HBV-DNA, ALT, AST, PLTs, PT, bilirubin; HCV variables: HCV-RNA, HCV genotype, ALT, AST, albumin, PLTs, PT, bilirubin. In Cohort C, the exploratory analyses in Long Covid patients include protein C reactive (PCR), D-Dimer levels, lymphocyte subpopulations (CD4+, CD8+, CD4/CD8, CD57+), interleukin 1, 6 and 8 and IFNy.
  Another exploratory objective is represented by the objective response rate (ORR) in patients who don't demonstrate TRAEs grade 3 or 4 of nivolumab plus ipilimumab in combination with platinum-based chemotherapy. Translational researches are also planned, involving circulating and tissue biomarkers to assess the immunological and inflammatory tumor microenvironment. In particular, the plasma samples will be collected at different timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Ricerche Cliniche, Verona, Veneto/Verona, Italy

IPD SHARING:
Plan to Share IPD: No